CLINICAL TRIAL: NCT04529460
Title: Post Market Clinical Study of a Point of Care COVID-19 IgG-IgM Rapid Test in Healthy Volunteers
Brief Title: Healthy Volunteer COVID-19 Antibody Testing Study
Status: Withdrawn | Type: Observational
Why Stopped: Funding withdrawn
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 134035
Record Dates: First submitted 2020-08-26; First posted 2020-08-27 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Previously COVID-19 positive: Previously confirmed PCR positive for COVID-19 And/or positive COVID-19 antibody test in the past six months
  Interventions: Diagnostic Test: COVID-19 antibody point of care test kit
- Previously COVID19 negative: No previous symptoms of COVID-19
  Interventions: Diagnostic Test: COVID-19 antibody point of care test kit

INTERVENTIONS:
Diagnostic Test: COVID-19 antibody point of care test kit — A disponible point of care test that identifies the presence of antibodies to COVID-19

SUMMARY:
The need for large-scale testing for COVID-19 has been highlighted by both the World Health Organization (WHO) and the UK government.

Immunity to coronavirus 2019 (COVID-19) infection can be determined by detecting the presence of antibodies to the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Immunoglobulins (Ig) to the SARS-CoV-2 develop during the second and third week of COVID-19 disease and can be detected by analyses conducted using laboratory tests. Accurate and scalable point-of-care testing (POCT) for the diagnosis of COVID-19 immunity would allow community diagnostic to be upscaled enormously. POCT for COVID-19 antibodies is possible using small disposable kits. POCT immunity testing using disposable kits will be imperative for effective surveillance and vaccinations programmes.

The study aims to test a novel, rapid antibody testing kit (IgG and IgM) in order to confirm its accuracy in a healthy volunteer population. The antibody testing kit intended for use in the study has already been CE marked for this purpose.

DETAILED DESCRIPTION:
This is a commercially funded prospective observational, cohort study of healthy volunteers to assess the sensitivity and specificity of a point of care antibody assay for COVID-19 (the ARIA COVID-19 IgG/IgM Rapid Test. The test is a disposable lateral flow chromatographic cassette (CTK Biotech, Inc., USA). The kit is CE approved for its intended purpose.

200 healthy volunteers will be enrolled into one of two cohorts:100 who have been confirmed to have had COVID-19 in the past (either by previous positive PCR swab or positive antibody test) and 100 thought not to have been affected by COVID-19. Once they have provided written informed consent to participate, volunteers will be invited to attend a 30 minutes appointment for testing. Prior to testing they will be asked to complete a short questionnaire to collect demographic information and details about previous symptoms of COVID-19.

A finger prick blood sample will be taken from the patient and then tested in the ARIA antibody kit. Afterwards, a routine blood sample (10 ml) will then be taken from the participant. The blood sample will be used in three separate ways:

1. A small sample of blood will be immediately removed from the sample bottle and placed into an ARIA antibody test kit.
2. One blood tube will be immediately centrifuged and a sample of plasma removed for use in the ARIA antibody testing kit.
3. One tube will be sent to the designated laboratory for formal COVID-19 ELISA antibody testing.

The ARIA antibody kit will be used to identify the presence of COVID-19 antibodies. The results will be compared to a laboratory enzyme-linked immunosorbent assay (ELISA) for COVID-19 antibodies. Once samples have arrived at the designated study laboratory they will undergo a specified ELSIA test for COVID-19 antibodies conducted according to the laboratory standard operating procedure for that test. For each sample type analysed (finger prick blood, venous blood, and plasma) the sensitivity and specificity of the test will be calculated against the results of the laboratory ELISA test.

Afterwards a brief exit questionnaire will be completed by the participant to document their experience of the study.

Recruitment is expected to be completed within six months of commencing the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged ≥ 18 years) healthy volunteers.
* For the positive group: PCR confirmed COVID-19 infection and/or positive antibodies test in the past six months,
* For the negative group: Never had symptoms of COVID-19
* Able to attend hospital for a blood and finger-prick test

Exclusion Criteria:

* Current symptoms of COVID-19
* Positive COVID-19 test result in the last 14 days
* Receiving or have received immunosuppression (including systemic corticosteroids) in the last 12 months
* Children (aged < 18years)
* Pregnancy
* Prisoners

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-01-29 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the COVID-19 antibody testing kit | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Martin, MB ChB, Principal Investigator — Royal Free Hospital NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No